CLINICAL TRIAL: NCT03411304
Title: Aortic Stenosis: Determinants and Prognostic Value of Preoperative Left Ventricular Remodeling After Valvular Replacement (AS-INTERVENTION)
Brief Title: Aortic Stenosis: Determinants and Prognostic Value of Preoperative Left Ventricular Remodeling After Valvular Replacement
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/080/HP
Record Dates: First submitted 2017-08-21; First posted 2018-01-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic valvular replacement; Aortic stenosis; Left ventricular remodeling; biomarkers
MeSH Terms: conditions — Aortic Valve Stenosis; Ventricular Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Aortic stenosis (AS) is the most frequent valvulopathy in Western countries. The prevalence of AS is constantly increasing due to the aging of the population. Although significant progress has been made in understanding the pathophysiological mechanisms underlying the onset and progression of AS, there is no medical treatment to slow or prevent its progression. The only treatment available is Aortic Valve Replacement (AVR) performed by surgery or by catheterization (TAVI).

AS is associated with an increase of post-load which leads the left ventricular myocardium to hypertrophy. Associated with hypertrophy, myocardial fibrosis will gradually develop. Despite interesting data, many unknowns persist and remain to be identified.

The aim of the study is to characterize prospectively the left ventricular remodeling and assess its changes after AVR and within 1 year in 500 patients using clinical, biological, echocardiographic and MRI parameters.

ELIGIBILITY:
Inclusion Criteria:

* Aortic stenosis
* Indication of Aortic Valve Replacement (Surgery or TAVI)

Exclusion Criteria:

* Rheumatismal or congenital aortic stenosis
* Aortic insufficiency (grade >= 2/4)
* Associated valvulopathy (grade >= 2/4)
* Myocardial infarction antecedent
* Severe renal failure
* Cardiac surgery (Aorta abdominal) antecedent
* Complex congenital cardiopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with at least moderate aortic stenosis and in whom an intervention is programmed or indicated
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of clinical events according to left ventricular remodeling | Year 1
  Echocardiography and MRI
Occurrence of clinical events according to left ventricular remodeling | Year 2
  Echocardiography and MRI
Occurrence of clinical events according to left ventricular remodeling | Year 3
  Echocardiography and MRI
Occurrence of clinical events according to left ventricular remodeling | Year 4
  Echocardiography and MRI

SECONDARY OUTCOMES:
Evolution of left ventricular remodeling after aortic valvular replacement | Year 1
  Echocardiography and MRI
Prognostic value of persistence and type of left ventricular remodeling | Year 1
  Echocardiography and MRI Occurence of clinical events
Prognostic value of fibrosis | Year 1
  Echocardiography and MRI Occurence of clinical events
Prognostic value of biomarkers | Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Helene Eltchaninoff, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- UH Rouen, Rouen, France